CLINICAL TRIAL: NCT03988517
Title: A Prospective Study Comparing Two-time Points of Thyroid Hormone Replacement During the Holy Month of Ramadan
Brief Title: Comparing Two-time Points of Thyroid Hormone Replacement During the Holy Month of Ramadan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. ZEINAB DABBOUS, Consultant Endocrine, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDABBOUS
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Hypothyroidism
Keywords: fasting
MeSH Terms: conditions — Hypothyroidism; Fasting

STUDY DESIGN:
Intervention Model Description: patients were block randomized into two groups according to the time they are going to take the leovthyroxine tablet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- levothyroxine at Iftar (Active Comparator): Patients took levothyroxine 30 minutes before breaking the fast at sunset (iftar)
  Interventions: Other: timing of receiving the drug
- Levothyroxine at Suhour (Active Comparator): Patients took levothyroxine 30 minutes before an early morning meal before sunrise (suhour)
  Interventions: Other: timing of receiving the drug

INTERVENTIONS:
Other: timing of receiving the drug — each group took levothyroxine in different timing

SUMMARY:
Muslims all over the world fast during the month of Ramadan from dawn until dusk. There is little data regarding the best timing of levothyroxine intake during the month of Ramadan where taking it on an empty stomach represents a challenge to most patients.This study aims to compare two-time points of levothyroxine intake during Ramadan in terms of change in thyroid stimulating hormone (TSH), compliance and convenience.

DETAILED DESCRIPTION:
Hypothyroidism requires regular replacement with levothyroxine to achieve euthyroidism (thyroid hormone status within the normal range). Usually, levothyroxine is taken orally in the morning on a daily basis. In clinical practice, the investigators have observed that this levothyroxine replacement is sub-optimal resulting in higher levels of thyroid stimulating hormone. Based on this observation, the investigators conducted this study to examine whether timing of oral intake of levothyroxine during the holy month of Ramadan will affect achievement of euthyroidism. They recruited 96 hypothyroid patients taking levothyroxine, attending Hamad endocrine outpatient clinics, who were fasting during Ramadan( May-June 2017)and for whom there is no clinical contraindication to fasting. Patients were randomly assigned to two time points for taking levothyroxine:

A. 30 minutes before the Iftar meal B. 30 minutes before Suhour The primary outcome was the change in thyroid stimulating hormone (TSH) before and after Ramadan. The null hypothesis is that there is no difference in TSH between the two groups.

The findings from the study will help in the clinical care of patients with hypothyroidism in Ramadan. Hypothyroidism is common worldwide and many Muslims will require the appropriate advice regarding management of hypothyroidism in Ramadan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Primary hypothyroidism who had stable TSH over the last 6 months prior to the study period
* Age between 18-70 years old
* Patients who planned to fast during Ramadan.

Exclusion Criteria:

* Patients with any end organ damage
* Pregnant ladies
* Patients with thyroid cancer
* Patients not adhering to medications
* Patients who had a clinical contraindication to observe fasting.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Change in TSH level | 1 month
  To evaluate the change in TSH level before and after Ramadan in the two groups.

SECONDARY OUTCOMES:
convenience and compliance | 1 month
  To determine in each group if the timing of levothyroxine dose was convenient and check the compliance with instructions to take levothyroxine in the assigned time. Done through clinical interview

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Abu Haliqa, MD, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad General Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data, but can provide them for researchers who ask for it